CLINICAL TRIAL: NCT02543710
Title: Biomarker Guided Treatment in Gynaecological Cancer
Acronym: Momatec2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/548
Record Dates: First submitted 2015-07-07; First posted 2015-09-07 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- phase 4 implementation study (Experimental): The historical MoMaTEC1 outcome data, collected from 2001-2015 serve as control arm. These data have been rigorously collected and quality controlled with extensive clinical annotation and follow-up data, and reflect the outcome in (for a larger part) the same population as expected for MoMaTEC2 as there have not been major changes in surgical or medical treatment for endometrial cancer in this time period that could cause confounding. Internal validity, and to a degree also external validity, covering practice in multiple countries, should in this way be assured.
  Interventions: Procedure: Biomarker (ER/PR) guided lymphadenectomy
- phase 2b biomarker study (Experimental): For the current study, stathmin is used as an integrated marker and does not dictate treatment modality, therefore there is no requirement for a control arm.
  Interventions: Drug: Biomarker guided weekly taxane treatment in endometrial/ ovarian cancer

INTERVENTIONS:
Procedure: Biomarker (ER/PR) guided lymphadenectomy — Lymphadenectomy in the pelvis and para-aortic, will, for patients who are considered otherwise low risk (endometrioid tumours grade 1 or 2, or grade 3 with <50% myometrial infiltration (MI), with no sign of extrauterine disease), be dependent on the preoperative hormone receptor status (ER and PR).
  Patients will be defined low risk when endometrioid, grade 1 or 2, or grade 3 with <50% MI, AND positive hormone receptor status for both ER AND PR. These patients will not undergo lymphadenectomy.
  Patients with endometrioid tumours grade 1 or 2, or grade 3 <50% MI,, with either negative ER or PR status, are defined high risk and will undergo pelvic and para-aortic lymphadenectomy as part of their surgical procedure.
  Patients will receive routine clinical follow-up for 5 years. Follow-up data will be collected for the study, focusing on survival and recurrence of disease. All patients will, as part of the study fill out validated quality of life questionnaires (QoL) at follow-up.
  Arms: phase 4 implementation study
Drug: Biomarker guided weekly taxane treatment in endometrial/ ovarian cancer — A 5mm tissue biopsy will be analysed for stathmin level in the recurrence as well as urine and a second 5mm biopsy on termination of study participation. The second biopsy could help explain why patients have stopped responding to the treatment. Determination of stathmin level both from the tissue and the urine will take place at the pathology department. Stathmin serves as an integrated biomarker, which enables a central biomarker analysis at Haukeland university hospital. Stathmin level is defined as high with an immunohistochemical score 9 (max score). All other scores are considered low. Pre-treatment all patients undergo CT or MRI, maximum 1 month prior to treatment start.
  During treatment, urine and bloods will be collected every treatment cycle (weekly basis). Imaging will take place every 8 treatment cycles. Treatment will continue until disease progression.
  Arms: phase 2b biomarker study

SUMMARY:
MoMaTEC2 aims to test, in clinically oriented studies, the applicability of already identified and promising molecular biomarkers, to promote individualisation of treatment for patients with endometrial cancer. Predominantly, but not exclusively, such biomarkers have shown to be interesting in retrospective analysis of our large prospectively collected MoMaTEC1 series.

Part 1: Performance of a phase 4 implementation trial for optimised stratification of surgical treatment, specifically the performance of (para-aortic and pelvic) lymphadenectomy guided by validated biomarkers.

Part 2: Performance of a phase 2b clinical biomarker study to evaluate the predictive potential of the biomarker stathmin for taxane treatment response in endometrial and ovarian cancer. In this study stathmin will be used as integrated biomarker.

ELIGIBILITY:
Inclusion Criteria part 1:

All patients referred to a participating research centre with suspicion of or confirmed endometrial cancer.

Exclusion Criteria part 1:

1. Patients who do not have endometrial cancer
2. Patients who will or cannot give informed consent (including language barriers)
3. Patients <18 years of age
4. Patients who will not get surgical treatment for their endometrial cancer

Inclusion criteria part 2:

1. Patients with endometrial or epithelial ovarian cancer who following routine clinical guidelines are offered weekly taxane (paclitaxel) treatment. This will often be a third or fourth line treatment, i.e. patients with advanced disease.
2. Technical possibility to obtain a new tissue biopsy to determine stathmin level in the tumour recurrence.

Exclusion criteria part 2:

1. Patients not suffering from endometrial or epithelial ovarian cancer
2. Patients <18 years of age
3. Patients who do not agree to the proposed treatment or will receive (part of) the treatment in a non-participating centre
4. Patients who cannot or do not want to give informed consent (including language barriers)

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
number of recurrences after primary treatment | 5 year after diagnosis
  The percentage of lymphadenectomy can be reduced safely and significantly, from 70% (MoMaTEC1 study results) to 30% in the MoMaTEC2 study through a better risk stratification of patients, especially better identification of low risk patients. Additionally The percentage of patients who need to be subjected to adjuvant (chemo) therapy can be reduced similarly from 20 to 10%, based on the same, optimised risk stratification and better identification of low risk patients. Patients will be rigorously followed during 5 years to detect any unexpected increase in the percentage of patients suffering a recurrence compared to the historical MoMaTEC1 cohort.
stathmin levels | duration of complete or partial treatment response in metastatic setting (expected duration less than one year)
  stathmin level will be measured in metastatic tissue and related to response to treatment using Response Evaluation Criteria In Solid Tumors (RECIST) criteria

SECONDARY OUTCOMES:
Quality of life measurements | 5 years post treatment
  Quality of life will be measured through validated questionnaires (EORTC QLQ-C30 and EORTC QLQ-EN24).
correlation of stathmin llevels in tumor, urine and blood | duration of complete or partial treatment response in metastatic setting (expected duration less than one year)
  stathmin tumor levels, urine levels and blood levels will be correlated.

CONTACTS AND LOCATIONS:
Overall Officials: Henrica MJ Werner, MD PhD MRCOG, Principal Investigator — Haukeland University Hospital
Locations (9):
- Radboud university hospital, Nijmegen, Netherlands
- Norway (7):
  - Women's hospital, Haukeland university hospital, Bergen, Hordaland
  - Ålesund hospital, Ålesund
  - Førde central hospital, Førde
  - Sørlandet hospital, Kristiansand
  - Akershus University hospital, Oslo
  - Stavanger university hospital, Stavanger
  - St Olav university hospital, Trondheim
- Spsk No 1, Lublin, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Forsse D, Barbero ML, Werner HMJ, Woie K, Nordskar N, Berge Nilsen E, Ellstrom Engh M, Vistad I, Rege A, Saevik-Lode M, Andreasen S, Haldorsen IS, Trovik J, Krakstad C. Longitudinal effects of adjuvant chemotherapy and lymph node staging on patient-reported outcomes in endometrial cancer survivors: a prospective cohort study. Am J Obstet Gynecol. 2022 Jan;226(1):90.e1-90.e20. doi: 10.1016/j.ajog.2021.08.011. Epub 2021 Aug 13. PMID 34400137